CLINICAL TRIAL: NCT04591613
Title: Late Clinical Events Associated With COVID-19 Infection: Multicenter Cohort
Brief Title: Late Clinical Events Associated With COVID-19 Infection
Acronym: COCO-LATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tourcoing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RIPH_2020_09
Record Dates: First submitted 2020-10-10; First posted 2020-10-19 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standardized clinical and paraclinical follow-up (Other): Standardized clinical and paraclinical follow-up will be offered in one of the referring investigator centers. Patients will be able to benefit from additional biological samples. Questionnaires will be completed by the patient or with the help of clinical research staff in paper format.
  All patients will make an inclusion visit (IV), then a clinical follow-up will be organized for the study at M4, M6, M12 from the day of the onset of the 1st symptoms of COVID.
  Quality of life and chronic disease impact scales will be completed at inclusion and follow-up visits.
  Total serum, plasma and naso-paaryngeal samples will be collected.
  Interventions: Other: Questionnaire; Other: Biocollection; Other: Follow-up visit

INTERVENTIONS:
Other: Questionnaire — Quality of life and chronic disease impact scales will be completed at inclusion and follow-up visits.
Other: Biocollection — Total serum, plasma samples will be collected
Other: Follow-up visit — All patients will make an inclusion visit (IV), then a clinical follow-up will be organized for the study at M4, M6, M12 from the day of the onset of the 1st symptoms of COVID.

SUMMARY:
Several publications document the occurrence of symptoms that persist or occur late.

The identification of the observed clinical manifestations and their clinical and paraclinical description are essential to better understand the natural evolution of COVID-19, to clarify the pathophysiological mechanism of these possible late manifestations, and to identify potential management options for patients.

Since this type of event is infrequent, a large-scale national multicenter cohort study focusing on symptomatic patients is needed.

DETAILED DESCRIPTION:
Several publications document the occurrence of symptoms that persist or occur late, more than 3 weeks after the first clinical manifestations of an SARS-COV2 infection. These manifestations may be related to thromboembolic or inflammatory complications, superinfections, or other mechanisms not yet well understood, including potentially related to the persistence of SARS-COV2. The identification of the observed clinical manifestations and their clinical and paraclinical description are essential to better understand the natural evolution of COVID-19, to clarify the pathophysiological mechanism of these possible late manifestations, and to identify potential management options for patients.

Since this type of event is infrequent, a large-scale national multicenter cohort study focusing on symptomatic patients is needed. In parallel, the prevalence of the main symptoms observed more than 3 weeks after the onset of a COVID-19 will be estimated through partnerships with existing cohort studies in the general population or in the population followed for COVID-19, still symptomatic or not at 3 weeks of infection.

Longitudinal implementation of bio-libraries will allow this cohort to also constitute a bridge between clinicians and researchers.

ELIGIBILITY:
Inclusion Criteria:

* History of symptomatic CoV-2-SARS infection as defined by :

  o Positive RT-PCR SARS-CoV-2 RT-PCR result OR positive SARS-CoV-2 serology

  o Associated with at least one event : x Anosmia occurring after February 2020 x OR COVID 19 evocative scanner x OR ≥ 2 contemporary symptoms of the virological sample from: asthenia, cough, dyspnea, fever, myalgia, dysgeusia, diarrhea AND not present prior to diagnosis
* AND persistence of at least one symptom present in the first 3 weeks of a COVID-19, more than 8 weeks away from the first symptoms of COVID-19. OR late onset of at least one new symptom a minimum of 3 weeks and a maximum of 6 months after the first symptoms of a CoV-2 SARS infection.
* First symptoms less than 6 months old on the day of inclusion
* To benefit from a State Health Insurance or Medical Aid plan
* Have signed an informed consent for inclusion.

Exclusion Criteria:

* Minor patient
* Patient under protection of justice
* Patient who required intensive care management :

  * more than 5 days
  * OR requiring orotracheal intubation
  * OR having required high flow ventilation (optiflow)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-12-31 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Clinical description of asthenia | At the end od the study, an average of 22 months
  Describe the frequence of asthenia between its onset and its disappearance. Assessment at baseline, then 4, 6 and 12 months.
Clinical description of dyspnea | At the end od the study, an average of 22 months
  Frequence of dyspnea between its onset and its disappearance. Assessment at baseline, then 4, 6 and 12 months. Assessment at baseline, then 4, 6 and 12 months.
Clinical description of thoracic disorders | At the end od the study, an average of 22 months
  Frequence of thoracic disorders between its onset and its disappearance. Assessment at baseline, then 4, 6 and 12 months. Assessment at baseline, then 4, 6 and 12 months.
Clinical description of neurological disorders | At the end od the study, an average of 22 months
  Frequence of neurological disorders between its onset and its disappearance. Assessment at baseline, then 4, 6 and 12 months. Assessment at baseline, then 4, 6 and 12 months.
Clinical description of anosmia | At the end od the study, an average of 22 months
  Frequence of anosmia disorders between its onset and its disappearance. Assessment at baseline, then 4, 6 and 12 months. Assessment at baseline, then 4, 6 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier ROBINEAU, MD PhD, Principal Investigator — CH TOURCOING
Locations (12):
- France (11):
  - Ch Auxerre, Auxerre
  - CHU Caen, Caen
  - CHRU Lille, Lille
  - CH Melun Marc Jacquet, Melun
  - CH Sud Seine et Marne, Nemours
  - AP-HP Hôpital Hôtel-Dieu, Paris
  - CHU de Saint-Etienne, Saint-Priest-en-Jarez
  - CH Tourcoing, Tourcoing
  - CHRU Tours, Tours
  - CHRU Nancy, Vandœuvre-lès-Nancy
  - Centre Hospitalier Bretagne Atlantique, Vannes
- CH André Rosemon de Cayenne, Cayenne, French Guiana

IPD SHARING:
Plan to Share IPD: No